CLINICAL TRIAL: NCT04399395
Title: Treatment With Naltrexone/Buprpion (Mysimba) to Optimize Weight Outcomes After Bariatric Surgery
Brief Title: Naltrexone/Bupropion (Mysimba) to Optimize Weight Outcomes After Obesity Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Covid-pandemic
Sponsor: Oslo University Hospital (Other)
Collaborators: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Principal Investigator, Serena Tonstad, Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32772
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Naltrexone; Bupropion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle and naltrexone/bupropion (Active Comparator)
  Interventions: Drug: Naltrexone/bupropion; Other: Lifestyle
- Lifestyle (Other)
  Interventions: Other: Lifestyle

INTERVENTIONS:
Drug: Naltrexone/bupropion — Approved drug for obesity treatment
  Arms: Lifestyle and naltrexone/bupropion
Other: Lifestyle — Lifestyle

SUMMARY:
Limited/poor weight loss and weight regain are concerns following bariatric surgery, and weight regain may increase the risk for relapse of comorbidities related to obesity. Medications for weight reduction may assist further weight loss, and support weight maintenance, with positive effects on comorbidities. This pilot study will examine the effect of naltrexone/bupropion and lifestyle advice versus lifestyle advice alone for 7 months in patients with a suboptimal weight trajectory (either little weight loss or weight regain) 2 years or later following bariatric surgery.

DETAILED DESCRIPTION:
Study aim and endpoints The aim of this pilot study is to evaluate the effect of Mysimba in patients with suboptimal weight loss or weight regain after bariatric surgery. The primary endpoint is body weight.

Objective The study objective is to understand whether patients with suboptimal weight loss or weight regain 2 years or more following bariatric surgery achieve better weight loss with Mysimba and dietary counselling compared with a control group treated with dietary counselling alone.

This is a phase IV, open label randomized controlled study conducted over 7 months with a 3-month post-intervention follow-up. The study will be conducted in accordance with good clinical practice. Patients meeting eligibility criteria will be randomized into one of two groups: an intervention group treated with Mysimba and lifestyle and a control group treated with lifestyle. The intervention group will be prescribed Mysimba gradually titrated to the maximum tolerated dose (maximum dose is 32 mg/360 mg divided in 4 tablets) with 2 week intervals. Both groups will receive the same follow up including dietary counselling during the course of the study. Randomization will be done using a standard internet-based program where group assignment cannot be anticipated. The study is not blinded.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 18-65 years who have undergone RYGB, mini-RYGB or sleeve gastrectomy 2 or more years previously and either

1. Have a percent total weight loss from time of surgery of <20% OR
2. Have a regain of at least 5% or more of nadir weight (lowest weight at 12-18 months after surgery) AND
3. Meet current clinical criteria for use of Mysimba (BMI ≥30 kg/m2 or BMI ≥27 kg/m2 with obesity-related comorbidity (diabetes type 2, controlled hypertension, dyslipidemia)

Exclusion Criteria:

* Serious illness or complications due to bariatric surgery according to the judgement of the investigators and clinical records
* Use of any weight loss medications following bariatric surgery
* Pregnancy or breastfeeding
* Participation in other weight loss studies
* Contraindication for use of Mysimba. These include but are not limited to epilepsy or history of seizure, uncontrolled hypertension (blood pressure ≥150/95 mmHg with or without medication), previous or current eating disorder, substance abuse, bipolar depression, serious liver or kidney disease, use of certain medications)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | 7 months
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Serena Tonstad, MD PhD, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No